CLINICAL TRIAL: NCT07140016
Title: A Phase 1b Study of Gilteritinib in Participants With Locally Advanced or Metastatic NSCLC With ALK Rearrangement After Prior Treatment With an ALK Inhibitor
Brief Title: A Study of Gilteritinib in Adults With Advanced ALK-positive Non-small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2215-CL-5201; 2025-522398-12 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-08-05; First posted 2025-08-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Anaplastic Lymphoma Kinase (ALK) Positive
Keywords: Non-small cell lung cancer (NSCLC); Anaplastic Lymphoma Kinase (ALK) Positive; gilteritinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — gilteritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- gilteritinib (Experimental): Participants will receive gilteritinib once daily in a 28-day cycle. For participants who are tolerant and achieve stable disease after 2 scans, a dose increase will be allowed.
  Interventions: Drug: gilteritinib

INTERVENTIONS:
Drug: gilteritinib — Oral
  Other Names: ASP2215

SUMMARY:
Genes give your body instructions on how to make proteins. Proteins are needed to keep the body working properly. Many types of cancer are caused by changes in certain genes, making them faulty. Some people with non small cell lung cancer (NSCLC) have a faulty ALK gene. ALK stands for anaplastic lymphoma kinase. People with NSCLC who have the faulty ALK gene are called ALK-positive. ALK inhibitors are an approved treatment for people with ALK positive NSCLC. Some people stop responding to treatment with ALK inhibitors over time due to more changes happening in their faulty ALK gene, so there is an unmet medical need. Gilteritinib is an approved treatment for people with acute myeloid leukemia (AML) with the faulty FLT3 gene who haven't responded to previous treatment, or their cancer came back after previous treatment. Gilteritinib also blocks changes in the ALK gene which could help people with ALK-positive NSCLC. A study needs to be done with gilteritinib in people with ALK-positive NSCLC.

The main aim of the study is to check the safety of gilteritinib in people with ALK-positive NSCLC and if they tolerate gilteritinib.

People in this study will be adults with locally advanced or metastatic ALK-positive non-small cell lung cancer (NSCLC). Locally advanced means the cancer has spread to nearby tissue. Metastatic means the cancer has spread to other parts of the body. They have stopped responding to treatment with ALK inhibitors, including alectinib or lorlatinib, over time. The key reasons people cannot take part are if they have symptomatic cancers in the brain or nervous system, their cancer has spread to the thin tissue that covers the brain and spinal cord (leptomengingeal metastasis), have recently had or planning to have major surgery, have certain heart conditions, or have recently had an infection, a stroke or mini-stroke.

People in the study will take tablets of gilteritinib once a day in a 28-day cycle. They may be given up to 2 different doses of gilteritinib. People in the study will start on the lower dose but can eventually switch to the higher dose if they tolerate the lower dose and meet the safety checks.

Whilst taking gilteritinib, people will have regular scans of their tumors. People will continue taking gilteritinib until their cancer gets worse, they have medical problems from gilteritinib that they can't tolerate, they ask to stop taking gilteritinib, they start other cancer treatment or, sadly pass away. People will visit the clinic about 7 days and then 30 days after they stop taking gilteritinib. They will be asked about any medical problems and will have a safety check. After this, people who stopped taking gilteritinib, but their cancer hadn't become worse, will continue to have regular scans of their tumors. If their cancer does get worse, they will no longer have scans of their tumors. After finishing gilteritinib, people will be phoned every 12 weeks to check on their health. People will be in the study for up to 4 years, depending on how they respond to gilteritinib.

ELIGIBILITY:
Inclusion Criteria:

* Participant has histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer (NSCLC) with a documented anaplastic lymphoma kinase (ALK) rearrangement and is not amenable to curative intent treatment.
* Participant is willing to submit, prior to enrollment, a fresh tumor tissue sample that was collected after completion of the most recent anti-cancer treatment and before the first dose of study intervention. If it is not medically feasible for a participant to provide a fresh tumor tissue sample, enrollment into the study should be confirmed with the Astellas medical monitor. In this case, an archival tumor tissue sample must be provided.
* Participant must have at least one prior line of ALK inhibitor-based therapy and meet one of the following criteria:

  * Participant received alectinib as the only prior ALK inhibitor regimen. Participant is eligible if chemotherapy was received in the neoadjuvant or adjuvant setting, and relapse or disease progressed after 12 months from completion of the treatment.
  * Participant received lorlatinib as one of the prior ALK inhibitor regimens.
* Participant has measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Participant has an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* Participant must have had progression or recurrence of NSCLC during or following receipt of the most recent therapy.
* Female participant is not pregnant and at least one of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP).
  * WOCBP who has a negative urine or serum pregnancy test within 7 days prior to the first dose of study intervention and agrees to follow the contraceptive guidance from the time of informed consent through at least 180 days after final study intervention administration.
* Female participant must not be breastfeeding or lactating starting at screening and throughout the investigational period and for 60 days after final study intervention administration.
* Female participant must not donate ova starting at the first administration of study intervention and throughout the investigational period and for 180 days after final study intervention administration.
* Male participant must agree to use contraception with female partner(s) of childbearing potential (including breastfeeding partner) throughout the treatment period and for 120 days after final study intervention administration.
* Male participant must agree to remain abstinent or use a condom with pregnant partner(s) for the duration of the pregnancy throughout the investigational period and for 120 days after final study intervention administration.
* Male participant must not donate sperm during the treatment period and for 120 days after final study intervention administration.
* Participant must meet the criteria as indicated on the clinical laboratory tests.
* Participant agrees not to participate in another interventional study while receiving study intervention in the present study/participating in the present study.

Exclusion Criteria:

* Participant has known oncogenic driver alterations other than ALK rearrangement.
* Participant has symptomatic central nervous system (CNS) metastases or has leptomeningeal metastasis.
* Participant has a history of malignancy other than NSCLC within 2 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix or malignancy considered cured with minimal risk of recurrence).
* Participant had major surgery (e.g., requiring general anesthesia) within 4 weeks prior to first dose of study intervention, or will not have fully recovered from surgery, or has surgery planned during the study treatment.
* Participant has ongoing clinically significant toxicity (Grade 2 or higher with the exception of alopecia) associated with prior anti-cancer treatment.
* Participant has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 28 days prior to first dose of study intervention.
* Participant has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease or a family history of long QT syndrome.
* Participant has a history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction or cardiac symptoms (including congestive heart failure) consistent with New York Heart Association Class III-IV within 6 months prior to the first dose of study intervention.
* Participant has a history of interstitial pneumonia.
* Participant had completed target therapy, radiotherapy, chemotherapy, biologics and/or immunotherapy within 14 days prior to first dose of study intervention.
* Participant requires treatment with strong inducers of cytochrome P450 (CYP) 3A.
* Participant requires treatment with concomitant drugs that target serotonin 5HT1 or 5HT2B receptors or sigma nonspecific receptor with the exception of drugs that are considered absolutely essential for the care of the participant.
* Participant has received any investigational therapy within 14 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has a mean Fridericia-corrected QT interval (QTcF) of > 450 msec at screening.
* Participant has known active hepatitis B virus (HBV) infection (defined as hepatitis B surface antigen (HBsAg)-positive and/or anti-HBV core antibody-positive) or known active hepatitis C virus (HCV) infection (defined as HCV RNA [qualitative] detected).

  * Participant with HBsAg-positivity and/or anti-HBV core antibody-positivity but with a negative HBV DNA PCR assay is permitted with appropriate antiviral prophylaxis or routine monitoring according to local practice.
  * Participant who has been curatively treated for HCV infection is permitted if he/she has documented sustained virologic response of 12 weeks.
* Participant has a known history of human immunodeficiency virus (HIV) infection with acquired immunodeficiency syndrome (AIDS)-related complications.
* Participant has echocardiogram (ECHO) or multigated acquisition scan (MUGA) at screening revealing left ventricular ejection fraction < 45%.
* Participant has any condition that makes the participant unsuitable for study participation.
* Participant has a known or suspected hypersensitivity to gilteritinib or any components of the formulation used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicity (DLT) | Up to 28 Days
  A Dose Limiting Toxicity is defined as any event meeting the DLT criteria occurring within 28 days of first dose.
Number of participants with Adverse Events (AEs) | Up to approximately 53 Months
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of participants with Serious Adverse Events (SAEs) | Up to approximately 53 Months
  An SAE is any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires hospitalization or prolongation to hospitalization, results in persistent or significant disability/incapacity, results in congenital anomaly or birth defect, or other medically important event.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to approximately 53 Months
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or adverse events (AEs) | Up to approximately 53 Months
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | Up to approximately 53 Months
  Number of participants with potentially clinically significant ECG values.
Number of participants with physical exam abnormalities and/or adverse events (AEs) | Up to approximately 53 Months
  Number of participants with potentially clinically significant physical exam values.
Number of participants at each grade of Eastern Cooperative Oncology Group (ECOG) performance status score | Up to approximately 53 Months
  The ECOG scale will be used to assess performance status. Grades range from 0 (fully active) to 5 (dead). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 53 Months
  ORR is defined as the proportion of participants whose best overall response is rated as confirmed Confirmed Response (CR) or Partial Response (PR) as assessed by investigator per Response Evaluation Criteria in Solid Tumors (RECIST) V1.1.
Duration of Response (DOR) | Up to approximately 53 Months
  DOR is defined as the time from the date of first documented response (CR or PR that is subsequently confirmed) to the date of first documented PD as assessed by investigator based on RECIST v 1.1. or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) | Up to approximately 53 Months
  DCR is defined as the proportion of participants whose best overall response is rated as confirmed CR, PR or stable disease as assessed by investigator based on RECIST v1.1.
Progression Free Survival (PFS) | Up to approximately 53 Months
  PFS is defined as the time from the date of first dose of study intervention until the date of first documented progressive disease (PD) as assessed by investigator based on RECIST v 1.1. or death due to any cause, whichever occurs first.
Intracranial Objective Response Rate (IC-ORR) | Up to approximately 53 Months
  IC-ORR is defined proportion of participants with intracranial lesions whose best overall response rate is rated as confirmed CR or PR as assessed by investigator based on RECIST v 1.1.
Overall Survival (OS) | Up to approximately 53 Months
  OS is defined as the time from the date of first dose of study intervention until the date of death from any cause.
Pharmacokinetics (PK) of gilteritinib in plasma: Concentration prior to dosing at multiple timepoints (Ctrough) | Up to approximately 6 Months
  Ctrough will be derived from the PK plasma samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development, Inc.
Locations (3):
- United States (3):
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Virginia Cancer Specialists PC, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Ou SI, Park CJ, Arter ZL, Nagasaka M. Successful and On-going Long-Term Disease Control (>24 Months) with Gilteritinib in an ALK+ NSCLC Patient with Brain Metastasis Who Has Progressed on Multiple ALK TKIs. A Case Report and Review of Literature on Gilteritnib. Lung Cancer (Auckl). 2025 Oct 22;16:139-145. doi: 10.2147/LCTT.S547128. eCollection 2025. PMID 41158152